CLINICAL TRIAL: NCT00790413
Title: High-dose MIBG With Subsequent Transplantation of Haploidentical Stem Cells in Children With Therapy Resistant Neuroblastoma
Brief Title: Haploidentical Stem Cell Transplantation in Neuroblastoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lund University Hospital (Other)
Responsible Party: Principal Investigator, Jacek Toporski, MD, PhD, Lund University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 385/2005
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Neuroblastoma
Keywords: Radiotherapy; Immunotherapy; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Neuroblastoma | interventions — 3-Iodobenzylguanidine; fludarabine; Thiotepa; Rituximab

ARMS (1):
- High-dose MIBG with haploidentical stem cell transplantation (Experimental): High-dose MIBG followed by Fludarabine, Thiotepa and Melfalan as conditioning Before haploidentical transplantation of T-cell depleted graft
  Interventions: Drug: iodine I 131 metaiodobenzylguanidine; Drug: Fludarabine; Drug: Thiotepa; Procedure: T-cell depletion; Procedure: Haploidentical stem cell transplantation; Procedure: Donor Lymphocyte Infusion; Drug: Rituximab; Procedure: Co-transplantation of mesenchymal stem cells

INTERVENTIONS:
Drug: iodine I 131 metaiodobenzylguanidine
Drug: Fludarabine
Drug: Thiotepa
Procedure: T-cell depletion
Procedure: Haploidentical stem cell transplantation
Procedure: Donor Lymphocyte Infusion
Drug: Rituximab
Procedure: Co-transplantation of mesenchymal stem cells

SUMMARY:
Children with primary resistant or relapsed neuroblastoma who do not achieve remission with conventional chemotherapy have extremely dismal prognosis. A novel treatment strategy combining tumor targeted radioisotope treatment with metaiodobenzylguanidine (MIBG) and immunotherapeutic effect of haploidentical stem cell transplantation (haploSCT) followed by low-dose donor lymphocyte infusions will be piloted. The use of the isotope is aimed to decrease pre-transplant tumour burden. Reduced intensity conditioning containing Fludarabine, Thiotepa and Melfalan will enable sustained engraftment as well as will serve as additional anti-tumor treatment. A prompt natural killer (NK)-cell mediated tumour control may be achieved by haploidentical stem cell transplantation. The investigators hypothesize that tumour cells potentially evading NK-cell mediated immunity may be targeted by infused donor T-cells and eliminated by either MHC-dependent manner or through a bystander effect. The possible graft versus tumor effect will be evaluated in children with therapy resistant neuroblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Refractory neuroblastoma (any chemo/radiosensitive stable disease)
* Relapse incl. autologous HSCT 3 m earlier
* Primary induction failure
* Cardiac output SF ≥25%
* Creatinine clearance ≥40 cc/min/1.73 m2
* Performance score of ≥50% (Lansky or Karnofsky)
* Available haploidentical family donor, aged ≥18 yrs, HIV-neg

Exclusion Criteria:

* Rapidly progressive disease
* Pregnancy

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2005-08; Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Engraftment rate | day 100

SECONDARY OUTCOMES:
Overall survival | 1 year
Immunological reconstitution | day 100
Incidence of acute graft versus host disease | day 100

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Toporski, MD, PhD, Principal Investigator — Lund University Hospital, Department of Pediatric Oncology
Locations (1):
- Lund University Hospital, Department of Pediatric Oncology and Bone Marrow Transplantation, Lund, Sweden

REFERENCES:
- [Background] Inoue M, Nakano T, Yoneda A, Nishikawa M, Nakayama M, Yumura-Yagi K, Sakata N, Yasui M, Okamura T, Kawa K. Graft-versus-tumor effect in a patient with advanced neuroblastoma who received HLA haplo-identical bone marrow transplantation. Bone Marrow Transplant. 2003 Jul;32(1):103-6. doi: 10.1038/sj.bmt.1704070. PMID 12815485
- [Background] Matthay KK, Tan JC, Villablanca JG, Yanik GA, Veatch J, Franc B, Twomey E, Horn B, Reynolds CP, Groshen S, Seeger RC, Maris JM. Phase I dose escalation of iodine-131-metaiodobenzylguanidine with myeloablative chemotherapy and autologous stem-cell transplantation in refractory neuroblastoma: a new approaches to Neuroblastoma Therapy Consortium Study. J Clin Oncol. 2006 Jan 20;24(3):500-6. doi: 10.1200/JCO.2005.03.6400. PMID 16421427
- [Background] Prigione I, Corrias MV, Airoldi I, Raffaghello L, Morandi F, Bocca P, Cocco C, Ferrone S, Pistoia V. Immunogenicity of human neuroblastoma. Ann N Y Acad Sci. 2004 Dec;1028:69-80. doi: 10.1196/annals.1322.008. PMID 15650233
- [Background] Neal ZC, Imboden M, Rakhmilevich AL, Kim KM, Hank JA, Surfus J, Dixon JR, Lode HN, Reisfeld RA, Gillies SD, Sondel PM. NXS2 murine neuroblastomas express increased levels of MHC class I antigens upon recurrence following NK-dependent immunotherapy. Cancer Immunol Immunother. 2004 Jan;53(1):41-52. doi: 10.1007/s00262-003-0435-2. Epub 2003 Sep 18. PMID 14504825
- [Background] Raffaghello L, Prigione I, Bocca P, Morandi F, Camoriano M, Gambini C, Wang X, Ferrone S, Pistoia V. Multiple defects of the antigen-processing machinery components in human neuroblastoma: immunotherapeutic implications. Oncogene. 2005 Jul 7;24(29):4634-44. doi: 10.1038/sj.onc.1208594. PMID 15897905
- [Background] Lang P, Pfeiffer M, Muller I, Schumm M, Ebinger M, Koscielniak E, Feuchtinger T, Foll J, Martin D, Handgretinger R. Haploidentical stem cell transplantation in patients with pediatric solid tumors: preliminary results of a pilot study and analysis of graft versus tumor effects. Klin Padiatr. 2006 Nov-Dec;218(6):321-6. doi: 10.1055/s-2006-942256. PMID 17080334
- [Result] Toporski J, Garkavij M, Tennvall J, Ora I, Gleisner KS, Dykes JH, Lenhoff S, Juliusson G, Scheding S, Turkiewicz D, Bekassy AN. High-dose iodine-131-metaiodobenzylguanidine with haploidentical stem cell transplantation and posttransplant immunotherapy in children with relapsed/refractory neuroblastoma. Biol Blood Marrow Transplant. 2009 Sep;15(9):1077-85. doi: 10.1016/j.bbmt.2009.05.007. Epub 2009 Jul 8. PMID 19660720
- [Result] Illhardt T, Toporski J, Feuchtinger T, Turkiewicz D, Teltschik HM, Ebinger M, Schwarze CP, Holzer U, Lode HN, Albert MH, Gruhn B, Urban C, Dykes JH, Teuffel O, Schumm M, Handgretinger R, Lang P. Haploidentical Stem Cell Transplantation for Refractory/Relapsed Neuroblastoma. Biol Blood Marrow Transplant. 2018 May;24(5):1005-1012. doi: 10.1016/j.bbmt.2017.12.805. Epub 2018 Jan 4. PMID 29307718